CLINICAL TRIAL: NCT04091867
Title: A Phase I/Ib Study of sEphB4-HSA in Combination With Chemotherapy or Cetuximab and Radiation Therapy in Patients With Intermediate to High Risk, Locally-Advanced Squamous Cell Carcinomas of the Head and Neck
Brief Title: sEphB4-HSA With RT+Chemo or Cetux in Patients With Intermediate to High Risk LAHNSCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Vasgene Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2575.cc; NCI-2019-06321 (Other: CTRP)
Record Dates: First submitted 2019-08-09; First posted 2019-09-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Cetuximab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This study will be enrolled using a 3+3 model. All patients will receive a fixed loading dose of 10 mg/kg to be followed by the assigned dose level during the concurrent phase. The 3+3 design model applies only to the concurrent phase. An expansion cohort of 6 patients will be added for testing biological endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sEphB4-HSA with CRT (Experimental): sEphB4-HSA: Loading dose at fixed dose of 10mg/Kg per below schema on D1 Concurrent dose per below schema D15-43 and given on an every other week basis Concurrent chemotherapy drug (either cisplatin or carboplatin): Per treating physician discretion, and treatment plan is based per NCCN guidelines. These can be administered in tri-weekly or weekly doses during the radiation period. The participant will receive the first infusion on Day 15 (+/- 3 days).
  Cetuximab:
  Loading dose 400 mg/m2 on D9 Concurrent dose 250mg/m2 weekly D15± 3 day window
  RT:
  6930 cGy IMRT starting D15-D18
  Interventions: Drug: sEphB4-HSA with chemotherapy; Drug: Cetuximab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: sEphB4-HSA with chemotherapy — sEphB4-HSA is a fusion protein combining the soluble extracellular EphB4 domain with albumin that targets the ephrin B2 receptor, which is thought to mediate resistance to EGFR-targeted therapy, and acts as a radiosensitizer by enhancing DNA damage and promoting apoptosis. Concurrent chemotherapy drug (either cisplatin or carboplatin): Per treating physician discretion, and treatment plan is based per NCCN guidelines. These can be administered in tri-weekly or weekly doses during the radiation period. The participant will receive the first infusion on Day 15 (+/- 3 days).
Drug: Cetuximab — Loading dose 400 mg/m2 on D9 Concurrent dose 250mg/m2 weekly D15± 3 day window
Radiation: Radiation Therapy — 6930 cGy IMRT starting D15-D18

SUMMARY:
This is a Phase I dose-escalation study of sEphB4-HSA in combination with chemotherapy, cetuximab and radiotherapy (RT). The purpose is to estimate the maximum tolerated dose (MTD) that can be administered concurrently with Cetuximab and radiation in patients with locally advanced, Stage III or IV A-B squamous cell carcinomas of the head or neck with a history of at least ten pack-years of smoking.

DETAILED DESCRIPTION:
RT combined with the EGFR-targeted agent cetuximab represents a valuable alternative to platinum-based CRT and is FDA-approved for initial treatment of LAHNSCC, but outcomes remain unfavorable. Recently, EphB4 has emerged as another rational target. While minimally expressed in normal tissue, it is highly expressed in LAHNSCC and has been implicated in resistance to both EGFR-targeted therapy and to RT. Suppression of EphB4 in the preclinical setting has enhanced tumor death and enhanced radiosensitivity. The novel agent sEphB4-HSA is a fusion protein that binds the ligand for EphB4 and leads to inhibition of tumor proliferation and angiogenesis. It was well-tolerated as monotherapy in a phase I trial but has yet to be explored in combination with radiotherapy or EGFR-directed treatments. A combined modality approach adding sEphB4-HSA to standard-of-care RT plus cetuximab represents a rational, targeted approach for investigation in patients with high risk LAHNSS p16-negative or any patient with heavy smoking histories. Moreover, a short window period of sEphB4-HSA monotherapy between baseline biopsy and repeat biopsy prior to initiation of cetuximab with RT will both minimize potential treatment delay and allow for the identification of potential biomarkers of response to sEphB4-HSA. Finally, a third optional biopsy, to be done if feasible after initiation of cetuximab-radiation, will allow us to identify radiosensitization markers and potential markers for treatment de-escalation. MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Patients must be willing to consent for two mandatory biopsies to be collected at baseline and again one week after the loading dose of sEphB4-HSA. A third optional biopsy will be collected if feasible 5-10 days after initiation of radiation treatment.
4. Be a male or female aged 18-100.
5. Pathologically confirmed (from the primary lesion and/or regional lymph nodes) squamous cell carcinoma of the oropharynx, hypopharynx, oral cavity, unknown primary, or larynx.
6. High risk, locally advanced HNSCC which may include any of the following by AJCC 8th Edition:

   * Stage III Hypopharyngeal Carcinoma AJCC v8
   * Stage III Laryngeal Cancer AJCC v8
   * Stage III Lip and Oral Cavity Cancer AJCC v8
   * Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8 or Stage III Oropharyngeal (p16-positive) Carcinoma ≥ 10 pack-years history of smoking
   * Stage IVA Hypopharyngeal Carcinoma AJCC v8
   * Stage IVA Laryngeal Cancer AJCC v8
   * Stage IVA Lip and Oral Cavity Cancer AJCC v8
   * Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8 or Stage IVA Oropharyngeal (p16-positive) Carcinoma ≥ 10 pack-years history of smoking
   * Stage IVB Hypopharyngeal Carcinoma AJCC v8
   * Stage IVB Laryngeal Cancer AJCC v8
   * Stage IVB Lip and Oral Cavity Cancer AJCC v8
   * Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8 or Stage IVB Oropharyngeal (p16-positive) Carcinoma ≥ 10 pack-years history of smoking
7. Patient is not a candidate for definitive surgical resection
8. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Total bilirubin < 1.5 x institutional upper limit of normal
   * AST and ALT < 2.5 x institutional upper limit of normal
9. For women of childbearing potential, a negative serum pregnancy test within 28 day screening to confirm eligibility. (Note: Pregnancy test will be repeated within 48 hours prior to the first dose of sEphB4-HAS) .
10. ECOG performance status ≤ 2.
11. Be deemed ineligible by a medical oncologist to receive concurrent platinum-based chemotherapy with radiotherapy or patient refusal of platinum-based chemotherapy.
12. Be deemed eligible by a medical oncologist to receive cetuximab.
13. Agreement to exercise appropriate use of contraception, as indicated.

    * For females of reproductive potential: use of highly effective contraception from time of screening through 12 weeks following the final dose of study treatment (see section 8.5).
    * For males of reproductive potential: use of condoms from time of screening through 12 weeks following the final dose of study treatment.
14. Pretreatment imaging to include the following within 28 days of treatment initiation:

    CT Neck (with contrast unless contraindicated) with CT chest OR PET-CT. MRI of the neck with contrast (unless contraindicated) can replace CT neck.

    N.B.: a CT Neck performed for radiation planning and read by a radiologist may serve as appropriate staging and planning tools.
15. General history and physical examination by a radiation or medical oncologist within 28 days prior to enrollment.
16. Examination by an ENT or head and neck surgeon, including laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) within 56 days prior to enrollment.
17. Dental evaluation and, if applicable, prophylaxis per NCCN guidelines performed within 84 days of treatment initiation.
18. Eligible for definitive therapy.

Exclusion Criteria:

1. Pregnant, attempting to conceive, lactating, or declining to use appropriate contraception for duration of study.
2. Hypertension that is uncontrolled (requiring 3+ antihypertensive medications to control).
3. Hypertension at screening (SBP ≥140mmHg or DBP ≥90mmHg, corresponding to Stage 2 according to JNC 7).
4. Prior history of allergic or infusion reaction to cetuximab or sEphB4.
5. Febrile illness within 7 days prior to enrollment.
6. Concomitant use of EGFR-directed therapies (besides cetuximab given as part of this trial), including erlotinib, gefitinib.
7. Major surgery (excluding tumor biopsy) within 4 weeks prior to start of study treatment.
8. Prior unrelated malignancy requiring current active treatment within 3 years prior to enrollment with exceptions of cervical carcinoma in situ, basal cell carcinoma of skin, resected T1-T2N0M0 differentiated thyroid cancers, Ta bladder cancer, prostatic adenocarcinoma of low or intermediate risk (per NCCN criteria).
9. Treatment with another investigational drug or other intervention within 30 days of treatment start.
10. Resectable oral cavity primary site
11. p16-positive carcinoma of the oropharynx or unknown primary that are T0-3, N0-1 (AJCC 8th Edition) AND ≤ 10 pack-year smoking history
12. Stage IVC (M1) disease per AJCC 8th edition.
13. Prior receipt of systemic chemotherapy for the study cancer (including "induction" or "neoadjuvant" chemotherapy) within 60 days of diagnosis; prior chemotherapy for a different cancer diagnosis is allowed.
14. Any severe, active comorbidity, defined as follows:

    * Cardiovascular disease or cerebrovascular disease, for example cerebrovascular accidents or myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or with the potential to interfere with protocol treatment;
    * Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to enrollment;
    * History or evidence upon physical/neurological examination of central nervous system disease (e.g., seizures) unrelated to cancer unless adequately controlled by medication;
    * Acute bacterial or fungal infection requiring intravenous antibiotics within 7 days of enrollment;
    * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
    * Patients known to be HIV positive or have active viral hepatitis, defined as positive HCV quantitative titers and/or +Hep B sAg and +IgM anti-HepB. Confirmatory testing is not required for the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is whether a dose-limiting toxicity (DLT) occurs | 13 weeks
  Severe cetuximab-associated rash is defined as per Lacouture 2010 criteria69, namely > 20 papules or pustules OR > 5 areas of erythema or edema < 1 cm (this is grade 3A) or > 20 papules/pustules OR > 5 areas of erythema or edema < 1 cm AND pain, pruritus, or effect on emotions or functioning (this is a commonly used criteria for grading of rash specifically related to EGFR inhibitors, such as cetuximab).

SECONDARY OUTCOMES:
To assess the effect of adding sEphB4-HSA to radiation and cetuximab in newly-diagnosed EGFR-expressing LAHNSCC and heavy smoking histories on Locoregional disease | 13 weeks
  Tumor response will be assessed in participants with measurable disease at start of therapy by measuring change in size (and/or FDG avidity) on CT (and/or PET/CT). LRC will be calculated as the time from completion of locoregional therapy until disease recurrence at the primary site or in the neck.
To assess the effect of adding sEphB4-HSA to radiation and cetuximab in newly-diagnosed EGFR-expressing LAHNSCC and heavy smoking histories on Distant Control | 13 weeks
  DC will be calculated as the time from completion of locoregional therapy until disease recurrence at a site other than the primary site or neck.
To assess the effect of adding sEphB4-HSA to radiation and cetuximab in newly-diagnosed EGFR-expressing LAHNSCC and heavy smoking histories on Disease Free Survival | 13 weeks
  DFS will be calculated as the time from completion of locoregional therapy until either disease recurrence at any site or until death.
Overall Survival | 13 weeks
  OS will be calculated as the time from diagnosis of LAHNSCC to death

OTHER OUTCOMES:
To assess target expression analysis, genomic, and immune analysis in tumor and blood samples obtained at baseline, after loading dose of s-EphB4-HSA, during CRT and at follow-up | 13 weeks
  To establish a gene signature panel on biopsy samples that can assess the response to sEphB4HSA
To assess target expression analysis, genomic, and immune analysis in tumor and blood samples obtained at baseline, after loading dose of s-EphB4-HSA, during CRT and at follow-up | 13 weeks
  Evaluate immune infiltration by multiplex immunofluorescence
To assess target expression analysis, genomic, and immune analysis in tumor and blood samples obtained at baseline, after loading dose of s-EphB4-HSA, during CRT and at follow-up | 13 weeks
  Blood samples to evaluate biomarkers of immune response including mass cytometry on circulating peripheral blood, and analysis of plasma cytokine, cleaved soluble ephrin-B2 as well as for evaluation of circulating auto-antibodies. Blood will be collected at baseline (before the administration of sEphB4) and after administration of sEphB4, as well as on day 22 of treatment and at the end of treatment at the follow-up visit. Cytokine mesoscale assays as well as Elisas will be used
To assess target expression analysis, genomic, and immune analysis in tumor and blood samples obtained at baseline, after loading dose of s-EphB4-HSA, during CRT and at follow-up | 13 weeks
  Tumor or nodal tissue taken at the time of initial biopsy and after sEphB4 HSA and will be profiled for whole gene and transcriptome sequencing of FFPE tissue, tumor infiltrating lymphocytes; activation markers and antigen specific TCR utilization/diversity.
To assess target expression analysis, genomic, and immune analysis in tumor and blood samples obtained at baseline, after loading dose of s-EphB4-HSA, during CRT and at follow-up | 13 weeks
  On long-term follow-up (6 months), tumor antigen specific T lymphocyte memory populations will be monitored for representation and robustness in in-vitro stimulation assays as potential biomarker of continued anti-tumor activity. PBMCs will be separately collected for this purpose.
To assess target expression analysis, genomic, and immune analysis in tumor and blood samples obtained at baseline, after loading dose of s-EphB4-HSA, during CRT and at follow-up | 13 weeks
  Circulating tumor DNA (ctDNA) will also be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No